CLINICAL TRIAL: NCT04155099
Title: Assessment of Cognitive Ability and the Intestinal Microbiome in Individuals With Liver Disease Before and After Investigational Microbiota Restoration Therapeutic
Brief Title: Investigational Microbiota Restoration Therapeutic for Hepatic Encephalopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Ochsner Health System (Other)
Collaborators: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019.193
Record Dates: First submitted 2019-08-21; First posted 2019-11-07 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver
Keywords: encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Study individuals will be placed into one of four study treatment groups: High dose investigational microbiota restoration therapeutic RBX7455 group, Low dose investigational microbiota restoration therapeutic RBX7455 group, or a pill quantity-matched Placebo group. Individuals will be randomized in a 1:1:1/2:1/2 manner. It is anticipated of the 75 potentially enrolled individuals, 50 will receive active treatment (high or low dose investigational microbiota restoration therapeutic) and 25 will receive placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study meaning both Ochsner study staff and participating individuals will not know to which group they are assigned/randomized. A third party will be responsible for providing study participant randomization and recording the exact treatment to which all study participants are assigned.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose (Experimental): Capsules of active drug will be supplied in 8-capsule blister packets to be taken twice per week for four weeks. Blood and stool samples and cognitive assessments will be collected before treatment and at 1, 3, 6, and 12 months after treatment.
  Interventions: Biological: RBX7455
- Low dose (Experimental): Capsules of active drug will be supplied in 4-capsule blister packets to be taken twice per week for four weeks. Blood and stool samples and cognitive assessments will be collected before treatment and at 1, 3, 6, and 12 months after treatment.
  Interventions: Biological: RBX7455
- pill quantity-matched Placebo (Placebo Comparator): Capsules of inactive compound will be supplied in 8- or 4-capsule blister packets to be taken twice per week for four weeks. Blood and stool samples and cognitive assessments will be collected before treatment and at 1, 3, 6, and 12 months after treatment.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RBX7455 — RBX7455 is a preparation of live intestinal microorganisms (active drug) purified from stool donations obtained from healthy, screened donors, mixed with preservative, lyophilized, and put into capsules. The capsules are taken orally (i.e., by mouth). After ingestion, these freeze-dried microorganisms can reconstitute and proliferate in the gut.
  Other Names: Microbiota Restoration Therapy
  Arms: High dose; Low dose
Biological: Placebo — Capsule with cellulose filler
  Arms: pill quantity-matched Placebo

SUMMARY:
Individuals with cirrhosis are likely to develop overt hepatic encephalopathy for which diagnostic modalities and treatment options are limited. The purpose of this study is to determine if individuals with cirrhosis who experience hepatic encephalopathy would benefit from investigational microbiota restoration therapy due to their inherent cognitive alterations. Analysis for a correlation between changes in microbiome composition and specific blood biomarkers could allow for earlier diagnosis of HE which could then be treated earlier and with novel treatments.

DETAILED DESCRIPTION:
The investigators hypothesize that changes in an individual's cognition due to HE-related liver cirrhosis can be stabilized and/or improved through investigational microbiota restoration therapeutic treatment. The main objective of this study is to determine if investigational microbiota restoration therapeutic treatment alters the cognitive function in individuals with cirrhosis who have been previously diagnosed with overt hepatic encephalopathy (HE). Once individuals have one HE episode, they are more likely to experience additional episodes, even after complying with standard of care. The number of HE episodes each study group experiences during the post-treatment follow-up will be compared among treatment groups. It is also anticipated that cognitive improvement will correlate with specific changes in the intestinal microbiota composition of these individuals likely shifting their microbiome away from baseline samples and becoming more like donor samples. Novel blood biomarkers potentially related to episodes of HE will be assessed in individuals before and after treatment.

ELIGIBILITY:
Inclusion Criteria

1. Individuals who are male or female and are between the ages of 18 and 70 years.
2. Individuals with a current diagnosis of liver cirrhosis as evidenced by one or more of the following:

   a. Liver Biopsy

   OR a clinical suspicion of cirrhosis based on the presence of one or more of the following criteria:
   1. Radiologic evidence of varices, cirrhosis or portal hypertension
   2. Laboratory evidence of platelet count <100,000 or AST/ALT ratio >1
   3. Endoscopic evidence of varices or portal gastropathy
   4. Elastography (i.e. Fibroscan)
3. Individuals must have at least one previously documented episode of HE.
4. Individuals must be able to read and write in the English language.
5. Individuals must be able and willing to utilize the electronic device necessary to measure cognitive function without assistance from outside individuals once the training phase has been completed.
6. Individuals must be able to provide valid informed consent prior to any study related procedures.

Exclusion Criteria

1. Individuals who are color-blind.
2. Individuals actively using psychotropic substances including alcohol.
3. Individuals who are pregnant, breastfeeding, or unwilling to practice birth control during participation in the study. Study individuals are expected to attest to this fact during their participation time. Females who are not surgically sterile or having undergone greater than one year of menopause will receive urine pregnancy tests at screening and initial drug dosing.
4. Presence of TIPS (transjugular intrahepatic portosystemic shunt).
5. Individuals with an active bacterial infection and are taking antibiotics for those infections at time of consent.
6. Individuals with ANC <800 (neutropenia).
7. Individuals with MELD >17.
8. Individuals with platelet count <35,000/mm3.
9. Individuals who are immunocompromised due any of the following reasons:

   1. HIV infection (CD4 count <200/mm3) or AIDS diagnosis
   2. Inherited/primary immunodeficiency disorders
   3. Treatment with any anti-neoplastic agent within the last 3 months (excluding locoregional therapy for hepatocellular carcinoma)
   4. Treatment with any immunosuppressant medications [including but not limited to monoclonal antibodies to B cells or T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil] within the last 3 months
10. Individuals who have previously undergone FMT.
11. Individuals with a history of colorectal cancer (all stages).
12. Individuals with a history of chronic intrinsic GI diseases such as inflammatory bowel disease (ulcerative colitis, Crohn's disease or microscopic colitis), eosinophilic gastroenteritis, celiac disease or irritable bowel syndrome as determined by Rome III criteria.
13. Individuals with a history of colectomy, major gastro-intestinal surgery, or intra-abdominal surgery.
14. Individuals with a history of Clostridium difficile infection six months prior to study enrollment.
15. Individuals with a history of chronic diarrhea.
16. Individuals currently participating in a research trial that involves drug or device intervention.
17. Individuals who are unable to fulfill all study criteria.
18. Individuals that the PI determines are not capable of participating in the research study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function at 1 month post-FMT as measured by change in response times on EncephalApp (Stroop test) | 1 month
  Determine whether microbiota restoration therapy improves cognition 1 month after treatment by measuring differences in time scores from EncephalApp. The app times participants in seconds (s) in variations of the Stroop Test. The average (s) across all trials will be reported as well as the difference in (s) between (trial 1)-(trial 5). Longer completion times indicate greater cognitive impairment, while a decrease in completion time from trial 1 to trial 5 indicates learning (cognitive improvement).
  The scale for this measure is theoretically 0s-500s.

SECONDARY OUTCOMES:
Number of HE episodes | 1 month to 12 months
  Once individuals have one HE episode, they are more likely to experience additional ones, even after complying with standard of care. The number of HE episodes each study group experiences during the post-treatment follow-up will be compared among treatment groups.
Engraftment of FMT as assessed by change in type and abundance of gut microbiota following shotgun sequencing | 1 month to 12 months
  It is anticipated that with treatment, changes in the intestinal microbiota composition of these individuals will likely shift their microbiome to contain different species. Microbiome analyses will measure, at the family and genus level, which bacteria are present and their relative abundance. Samples from the same individual at different time points will be compared as well as differences between treatment groups at each time point.
Change in cognitive function at 3, 6 and 12 months post-FMT as measured by change in response times on EncephalApp (Stroop test) | 3 to 12 months
  Determine whether microbiota restoration therapy improves cognition 3, 6, and 12 months after treatment by measuring differences in time scores from EncephalApp. The app times participants in seconds (s) in variations of the Stroop Test. The average (s) across all trials will be reported as well as the difference in (s) between (trial 1)-(trial 5). Longer completion times indicate greater cognitive impairment, while a decrease in completion time from trial 1 to trial 5 indicates learning (cognitive improvement).

OTHER OUTCOMES:
Correlations of clinical variables with primary and secondary outcomes | Duration of the study (0 days to 12 months)
  Other clinical outcome variables available from individuals' electronic medical records include age, liver-related diagnoses and disease progression, antibiotic usage history, number of previous hospitalizations, and mortality. This clinical data will be analyzed for significant correlations with the primary and secondary outcome variables.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Garcia-Diaz, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No